CLINICAL TRIAL: NCT03731455
Title: A Prospective, Interventional, Multi-center, Open-label, Premarket Study to Evaluate Safety, Performance and Usability of the Wise Cortical Strip for Intraoperative Neurophysiological Monitoring (WIN Study)
Brief Title: WISE Cortical Strip for Intraoperative Neurophysiological Monitoring
Acronym: WIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wise S.r.l. (Industry)
Collaborators: Genae (Industry); Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 001_WCS
Record Dates: First submitted 2018-10-30; First posted 2018-11-06 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Brain Tumor Adult; Epilepsy
Keywords: Cortical strip; Electrode
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: The neurosurgical intervention will be performed with both devices: investigational (Wise Cortical Strip, WCS) and comparator device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigational and Comparator devices (Experimental): Investigational (WISE Cortical Strip, WCS) and comparator (Subdural Strip Electrode, Ad-Tech Medical Instruments Corporation) devices will be used together.
  Interventions: Device: WISE Cortical Strip

INTERVENTIONS:
Device: WISE Cortical Strip — The WISE Cortical Strip is a medical device composed by a strip and by a cable.

SUMMARY:
The WIN Study is a prospective, interventional, multi-center, open-label premarket study designed to confirm the safety, performance and intended use of the WISE Cortical Strip (WCS) for CE certification purposes. Participants with documented diagnosis of epilepsy or brain tumor requiring intracranial surgery, who meet all eligibility criteria, will undergo IntraOperative Neurophysiological Monitoring (IONM) during a neurosurgical intervention with the WCS and a comparator device.

DETAILED DESCRIPTION:
The IONM is the use of electrophysiological methods to identify important neural structures in the operative field, including eloquent areas, in order to monitor their functional integrity during the neurosurgical lesion resection. The benefit of performing functional monitoring of the areas surrounding the lesion is to minimize neurological damages during surgical lesions resection and thus to avoid and/or limit significant post-operative impairments. During the therapeutic resection of brain tumors or epileptogenic lesions, the use of the IONM is associated to other intraoperative techniques (e.g. brain mapping techniques) that, together to combined efforts of a multidisciplinary team of neurosurgeons, neuroradiologists, neuropsychologists, and neurophysiologists, contribute to the definition of location, extension, and extent of functional involvement that a lesion causes in an individual participant.

The principal electrophysiological methods to perform the IONM are the recording of brain's electrical activities (Somatosensory Evoked Potentials, SEPs and ElectroCorticoGraphy, ECoG) and electrical stimulation of motor regions (to elicit Motor Evoked Potentials, MEPs) using cortical strips placed on surface of the brain.

Thus, the WCS is intended to be used intraoperatively on the brain surface, to perform brain monitoring.

ELIGIBILITY:
Inclusion criteria:

1. Brain tumor or epilepsy that require neurosurgical intervention and exposure of the central region of the cerebral cortex including at least the hand-forearm areas in the primary motor cortex and the primary somatosensory cortex (i.e. excision of lesion, open approach)
2. Age: 18 - 75 years at the time of enrollment
3. Required intraoperative neurophysiological monitoring with subdural electrodes
4. Willingness to provide informed consent for participating in the study

Exclusion critria:

1. Significant psychiatric impairments which, in the opinion of the investigator, will interfere with the proper administration or completion of the protocol
2. Acute or untreated infections (viral, bacterial or fungal)
3. Currently on any anticoagulant medication that cannot be discontinued during the perioperative period, or patients with factor XIII deficiency or any other hematological disease
4. Current treatment with antibiotics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Device Effects (SADEs) of the WISE Cortical Strip. | For the entire duration of the surgeries and after 24 hours
The Signal-to-Noise Ratio percentage (SNR%) calculated on Somatosensory Evoked Potential (SEP) signals. | During the surgery

SECONDARY OUTCOMES:
Impedance values measured for the WISE Cortical Strip. | During the surgery
Motor Evoked Potentials (MEPs). | During the surgery
Dedicated usability questionnaire. | Following surgeries

CONTACTS AND LOCATIONS:
Locations (5):
- Klinikum der Universitat München, Munich, Germany, Germany
- Azienda Ospedaliera Universitaria Integrata Verona (AOUI Verona), Verona, Verona, Italy
- Switzerland (3):
  - Inselspital, Bern, Switzerland
  - Luzerner Kantonsspital, Lucerne, Switzerland
  - Universitätsspital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fedele T, Schonenberger C, Curio G, Serra C, Krayenbuhl N, Sarnthein J. Intraoperative subdural low-noise EEG recording of the high frequency oscillation in the somatosensory evoked potential. Clin Neurophysiol. 2017 Oct;128(10):1851-1857. doi: 10.1016/j.clinph.2017.07.400. Epub 2017 Jul 27. PMID 28826015
- [Background] Kim SM, Kim SH, Seo DW, Lee KW. Intraoperative neurophysiologic monitoring: basic principles and recent update. J Korean Med Sci. 2013 Sep;28(9):1261-9. doi: 10.3346/jkms.2013.28.9.1261. Epub 2013 Aug 28. PMID 24015028
- [Background] Macdonald DB. Intraoperative motor evoked potential monitoring: overview and update. J Clin Monit Comput. 2006 Oct;20(5):347-77. doi: 10.1007/s10877-006-9033-0. Epub 2006 Jul 11. PMID 16832580
- [Background] Aungaroon G, Zea Vera A, Horn PS, Byars AW, Greiner HM, Tenney JR, Arthur TM, Crone NE, Holland KD, Mangano FT, Arya R. After-discharges and seizures during pediatric extra-operative electrical cortical stimulation functional brain mapping: Incidence, thresholds, and determinants. Clin Neurophysiol. 2017 Oct;128(10):2078-2086. doi: 10.1016/j.clinph.2017.06.259. Epub 2017 Jul 18. PMID 28778475